CLINICAL TRIAL: NCT05564039
Title: A Phase 4, Randomized, Open-Label, Active-Controlled Study to Investigate the Efficacy and Safety of Switching From Weekly Dulaglutide to Weekly Tirzepatide in Adults With Type 2 Diabetes
Brief Title: A Study of Tirzepatide (LY3298176) in Adult Participants With Type 2 Diabetes Switching From Dulaglutide (SURPASS-SWITCH)
Acronym: SURPASS-SWITCH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18395; I8F-MC-GPIH (Other: Eli Lilly and Company); 2022-500101-41-00 (Other: EU Trial Number)
Record Dates: First submitted 2022-09-30; First posted 2022-10-03 (Actual); Results first posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Tirzepatide; dulaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 15 Milligram (mg) Tirzepatide or Maximum Tolerated Dose (MTD) (Experimental): Participants received tirzepatide administered as subcutaneous (SC) injection via a single-dose pen (SDP) once weekly (QW) for 40 weeks.
  The starting dose of tirzepatide was 2.5 mg QW, which increased by 2.5 mg every 4 weeks (2.5 mg to 5 mg to 7.5 mg to 10 mg to 12.5mg to 15 mg) until 15 mg or MTD was reached.
  Interventions: Drug: Tirzepatide
- 4.5 mg Dulaglutide or MTD (Active Comparator): Participants received dulaglutide administered as SC injection via a SDP QW for 40 weeks.
  The starting dose of dulaglutide was either 1.5 mg QW, which increased by 1.5 mg every 4 weeks (1.5 mg to 3 mg to 4.5 mg) until 4.5 mg or MTD was reached, or 3.0 mg QW, which increased to 4.5 mg after 4 weeks or until MTD was reached.
  Interventions: Drug: Dulaglutide

INTERVENTIONS:
Drug: Tirzepatide — Administered SC
  Other Names: LY3298176
  Arms: 15 Milligram (mg) Tirzepatide or Maximum Tolerated Dose (MTD)
Drug: Dulaglutide — Administered SC
  Other Names: LY2189265
  Arms: 4.5 mg Dulaglutide or MTD

SUMMARY:
The main purpose of this study is to investigate the efficacy and safety of switching from weekly dulaglutide to weekly tirzepatide compared to increasing the dulaglutide dose in adults with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Have type 2 diabetes
* Have HbA1c ≥7.0% (≥53 mmol/mol) to ≤9.5% (≤80 mmol/mol)
* Are currently on a stable dose of dulaglutide weekly (0.75 mg or 1.5 mg) for at least 6 months prior to screening.
* No treatment with oral antihyperglycemic medication (OAM), or on a stable dose of up to 3 OAMs, which may include metformin, sodium glucose cotransporter-2 inhibitors (SGLT-2i), and/or sulfonylurea, for at least 3 months before screening.
* Have had stable body weight (±5%) during the 90 days preceding screening
* Have BMI ≥25 kilogram/square meter (kg/m²)

Exclusion Criteria:

* Have type 1 diabetes
* Have a history of chronic or acute pancreatitis
* Have a history of

  * proliferative diabetic retinopathy, or
  * diabetic maculopathy, or
  * nonproliferative diabetic retinopathy that requires acute treatment.
* Have any of these cardiovascular (CV) conditions within 60 days prior to screening:

  * acute myocardial infarction,
  * cerebrovascular accident (stroke), or
  * hospitalization due to congestive heart failure (CHF).
* Have New York Heart Assocation (NYHA) Functional Classification Class IV CHF
* Have family or personal history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN2).
* Have within 90 days prior to screening received treatment with medications intended to promote weight loss. This includes prescribed, over-the-counter, or alternative remedies
* Have an estimated glomerular filtration rate (eGFR) <30 mL/minute/1.73 m2 (or lower than the country-specific threshold for discontinuing metformin therapy per local label)
* Have been treated with insulin prior to screening

  * Exception: use of insulin for gestational diabetes or short-term use (<14 days) for acute conditions such as acute illness, hospitalization, or elective surgery.
* Have a history of reduction of dose of dulaglutide, due to intolerability, without successful reescalation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2022-11-30 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (36):
- United States (10):
  - ALL Medical Research, LLC, Cooper City, Florida
  - Metabolic Research Institute, Inc., West Palm Beach, Florida
  - NorthShore University Health System, Skokie, Illinois
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - Clinvest Research LLC, Springfield, Missouri
  - Alliance for Multispecialty Research, LLC, Norman, Oklahoma
  - Juno Research, Houston, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Southern Endocrinology Associates, Mesquite, Texas
  - North Hills Family Medicine/North Hills Medical Research, North Richland Hills, Texas
- Belgium (6):
  - Imelda General Hospital, Bonheiden, Antwerpen
  - Antwerp University Hospital, Edegem, Antwerpen
  - ZNA Jan Palfijn, Merksem, Flanders
  - AZ Nikolaas, Sint-Niklaas, Oost-Vlaanderen
  - UZ Leuven, Leuven, Vlaams-Brabant
  - Az Damiaan vzw, Ostend, West-Vlaanderen
- Germany (6):
  - InnoDiab Forschung Gmbh, Essen, North Rhine-Westphalia
  - Institut für Diabetesforschung GmbH Münster, Münster, North Rhine-Westphalia
  - Studienzentrum Dr. Tasso Bieler, Riesa, Saxony
  - RED-Institut GmbH, Oldenburg in Holstein, Schleswig-Holstein
  - Medizinisches Versorgungszentrum am Bahnhof Spandau, Spandau, State of Berlin
  - Diabeteszentrum Hamburg West, Hamburg
- Mexico (8):
  - Diseno y Planeacion en Investigacion Medica, Guadalajara, Jalisco
  - Unidad de Investigación Clínica y Atención Médica HEPA, Guadalajara, Jalisco
  - Centro Especializado En Diabetes, Obesidad Y Prevencion De Enfermedades Cardiovasculares, Mexico City, Mexico City
  - Instituto de Diabetes, Obesidad y Nutricion, Cuernavaca, Morelos
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León
  - Unidad biomedica avanzada monterrey, Monterrey, Nuevo León
  - Centro de Estudios de Investigacion Metabolicos y Cardiovasculares, Ciudad Madero, Tamaulipas
  - Investigacion En Salud Y Metabolismo Sc, Chihuahua City
- Romania (6):
  - Diabdana, Oradea, Bihor County
  - Mariodiab Clinic, Brasov, Brașov County
  - Geea Medical Easy Diet, Bucharest, București
  - Gama Diamed, Mangalia, Constanța County
  - CMI DNBM Dr. Pop Lavinia, Baia Mare, Maramureş
  - Clinica Korall, Satu Mare

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Billings LK, Winne L, Sharma P, Gomez-Valderas E, Chivukula KK, Kwan AYM. Comparison of Dose Escalation Versus Switching to Tirzepatide Among People With Type 2 Diabetes Inadequately Controlled on Lower Doses of Dulaglutide : A Randomized Clinical Trial. Ann Intern Med. 2025 May;178(5):609-619. doi: 10.7326/ANNALS-24-03849. Epub 2025 Apr 4. PMID 40183678
- See also: A Study of Tirzepatide (LY3298176) in Adult Participants With Type 2 Diabetes Switching From Dulaglutide (SURPASS-SWITCH) — https://trials.lilly.com/en-US/trial/362875

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 15 Milligram (mg) Tirzepatide or Maximum Tolerated Dose (MTD) | 4.5 mg Dulaglutide or MTD
Started | 139 | 143
Received at Least 1 Dose of Study Drug | 139 | 143
Completed | 129 | 134
Not Completed | 10 | 9
Not completed — Adverse Event | 1 | 0
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 3 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Inadvertent enrollment | 3 | 6

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- 15 mg Tirzepatide or MTD: Participants received tirzepatide administered as SC injection via a SDP QW for 40 weeks.
  The starting dose of tirzepatide was 2.5 mg QW, which increased by 2.5 mg every 4 weeks (2.5 mg to 5 mg to 7.5 mg to 10 mg to 12.5 mg to 15 mg) until 15 mg or MTD was reached.
- Total: Total of all reporting groups
Arm/Group | 15 mg Tirzepatide or MTD | 4.5 mg Dulaglutide or MTD | Total
Number analyzed (Participants) | 139 | 143 | 282
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (9.8) | 57.3 (10.0) | 57.6 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 72 | 136
  Male | 75 | 71 | 146
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 14 | 32
  Not Hispanic or Latino | 18 | 19 | 37
  Unknown or Not Reported | 103 | 110 | 213
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 23 | 19 | 42
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 109 | 120 | 229
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 9 | 10 | 19
  Germany | 19 | 21 | 40
  Mexico | 43 | 48 | 91
  Romania | 32 | 31 | 63
  United States | 36 | 33 | 69
Percentage of Hemoglobin A1c (HbA1c) at Baseline [Mean (Standard Deviation); unit: Percentage of HbA1c] — HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time.
  Percentage of HbA1c | 7.82 (0.69) | 7.82 (0.73) | 7.82 (0.71)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c
Description: HbA1c is the glycated fraction of hemoglobin A. HbA1c is measured primarily to identify average plasma glucose concentration over prolonged periods of time. Least squares (LS) mean was calculated using mixed model repeated measures (MMRM) for post-baseline measures: Variable = Baseline + Number of Background OAMs Group 1 + Dulaglutide Dose at Screening + Geographic Region 1 + Treatment + Time + Treatment*Time (Type III sum of squares). Variance-Covariance structure (Actual Value) = Unstructured. Variance-Covariance structure (Change from Baseline) = Unstructured.
Time Frame: Baseline, Week 40
Population: All randomly assigned participants who took at least 1 dose of study drug and had a baseline and at least 1 post-baseline value for this outcome, excluding participants discontinuing study drug due to inadvertent enrollment and data after initiating rescue antihyperglycemic medication or prematurely stopping study drug.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | 15 mg Tirzepatide or MTD | 4.5 mg Dulaglutide or MTD
Number analyzed (Participants) | 114 | 105
percentage of HbA1c | -1.59 (0.073) | -0.69 (0.074)
Statistical Analysis 1: Comparison: 15 mg Tirzepatide or MTD vs 4.5 mg Dulaglutide or MTD; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean difference (Final Values) = -0.90, 95% CI 2-sided [-1.10 to -0.69]

2. Secondary Outcome: Change From Baseline in Body Weight
Description: LSMean was calculated using MMRM for post-baseline measures: Variable = Baseline + Number of Background OAMs Group 1 + Dulaglutide Dose at Screening + Geographic Region 1 + Baseline HbA1c Group + Treatment + Time + Treatment*Time (Type III sum of squares). Variance-Covariance structure (Actual Value) = Unstructured. Variance-Covariance structure (Change from Baseline) = Unstructured.
Time Frame: Baseline, Week 40
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kilograms (kg)
Arm/Group | 15 mg Tirzepatide or MTD | 4.5 mg Dulaglutide or MTD
Number analyzed (Participants) | 123 | 111
kilograms (kg) | -11.0 (0.48) | -3.6 (0.49)
Statistical Analysis 1: Comparison: 15 mg Tirzepatide or MTD vs 4.5 mg Dulaglutide or MTD; Test type: Superiority; p < .0001, Mixed Models Analysis; LS Mean difference (Final Values) = -7.4, 95% CI 2-sided [-8.7 to -6.0]

3. Secondary Outcome: Percentage of Participants Who Achieved HbA1c <7%
Description: The percentage of participants was calculated by dividing the number of participants reaching target HbA1c by the total number of participants analyzed, multiplied by 100. Analyses included all participants having non-missing baseline and at least one non-missing post-baseline value of the response variable. Missing endpoint measures are imputed by predictions from an MMRM analysis model using observed data in the efficacy analysis set and adjusted for Baseline HbA1c Value, Baseline SGLT2i use(Yes/No), Treatment, Visit, and Treatment by Visit interaction.
Time Frame: Week 40
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 15 mg Tirzepatide or MTD | 4.5 mg Dulaglutide or MTD
Number analyzed (Participants) | 114 | 105
percentage of participants | 84.21 | 52.38
Statistical Analysis 1: Comparison: 15 mg Tirzepatide or MTD vs 4.5 mg Dulaglutide or MTD; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 7.13, 95% CI 2-sided [3.82 to 13.32]

4. Secondary Outcome: Percentage of Participants Who Achieved HbA1c <=6.5%
Description: The percentage of participants was calculated by dividing the number of participants reaching target HbA1c by the total number of participants analyzed, multiplied by 100. Analyses included all participants having non-missing baseline and at least one non-missing post-baseline value of the response variable. Logistic regression model was used with missing endpoint measures imputed by predictions from an MMRM analysis model using observed data in the efficacy analysis set and adjusted for baseline HbA1c, geographic region 1, number of background OAMs in group 1, dulaglutide dose at screening, and treatment as factors.
Time Frame: Week 40
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 15 mg Tirzepatide or MTD | 4.5 mg Dulaglutide or MTD
Number analyzed (Participants) | 134 | 132
percentage of participants | 73.88 | 22.73
Statistical Analysis 1: Comparison: 15 mg Tirzepatide or MTD vs 4.5 mg Dulaglutide or MTD; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 12.24, 95% CI 2-sided [6.51 to 23.02]

5. Secondary Outcome: Percentage of Participants Who Achieved HbA1c <5.7%
Description: as for outcome 4
Time Frame: Week 40
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 15 mg Tirzepatide or MTD | 4.5 mg Dulaglutide or MTD
Number analyzed (Participants) | 134 | 132
percentage of participants | 21.64 | 2.27
Statistical Analysis 1: Comparison: 15 mg Tirzepatide or MTD vs 4.5 mg Dulaglutide or MTD; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 15.34, 95% CI 2-sided [4.58 to 51.36]

6. Secondary Outcome: Percentage of Participants Who Achieve Weight Loss From Baseline of ≥5%
Description: Missing endpoint measures are imputed by predictions using observed data in the efficacy analysis set from the same treatment group through an MMRM analysis model for post-baseline measures: Variable = Baseline + Geographic Region 1 + Number of Background OAMs Group 1 + Dulaglutide Dose at Screening + Baseline HBA1C Group + Treatment + Time + Treatment*Time.
Time Frame: Week 40
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 15 mg Tirzepatide or MTD | 4.5 mg Dulaglutide or MTD
Number analyzed (Participants) | 134 | 131
percentage of participants | 84.33 | 37.40
Statistical Analysis 1: Comparison: 15 mg Tirzepatide or MTD vs 4.5 mg Dulaglutide or MTD; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 9.31, 95% CI 2-sided [5.11 to 16.98]

7. Secondary Outcome: Percentage of Participants Who Achieve Weight Loss From Baseline of ≥10%
Description: as for outcome 6
Time Frame: Week 40
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 15 mg Tirzepatide or MTD | 4.5 mg Dulaglutide or MTD
Number analyzed (Participants) | 134 | 131
percentage of participants | 58.21 | 6.87
Statistical Analysis 1: Comparison: 15 mg Tirzepatide or MTD vs 4.5 mg Dulaglutide or MTD; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 19.35, 95% CI 2-sided [9.07 to 41.30]

8. Secondary Outcome: Percentage of Participants Who Achieve Weight Loss From Baseline of ≥15%
Description: as for outcome 6
Time Frame: Week 40
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 15 mg Tirzepatide or MTD | 4.5 mg Dulaglutide or MTD
Number analyzed (Participants) | 134 | 131
percentage of participants | 27.61 | 0.76
Statistical Analysis 1: Comparison: 15 mg Tirzepatide or MTD vs 4.5 mg Dulaglutide or MTD; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 35.83, 95% CI 2-sided [7.18 to 178.89]

9. Secondary Outcome: Percentage of Participants Who Achieved Composite Endpoint (HbA1c <=6.5% & Weight Loss >=10% & No-Hypoglycemia)
Description: A composite endpoint is defined as HbA1c ≤ 6.5%, weight loss ≥ 10%, and no hypoglycemia, defined as blood glucose (BG) <3.0 millimole/liter (mmol/L) and/or severe hypoglycemia. Missing endpoint measures are imputed by predictions using observed data in the efficacy analysis set from the same treatment group through an MMRM analysis model for post-baseline measures:
  For HbA1c: Variable = Baseline + Geographic Region 1 + Number of Background OAMs Group 1 + Dulaglutide Dose at Screening + Treatment + Time + Treatment*Time.
  For Weight: Variable = Baseline + Geographic Region 1 + Number of Background OAMs Group 1 + Dulaglutide Dose at Screening + Baseline HbA1c Group + Treatment + Time + Treatment*Time.
Time Frame: Week 40
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 15 mg Tirzepatide or MTD | 4.5 mg Dulaglutide or MTD
Number analyzed (Participants) | 133 | 131
percentage of participants | 46.62 | 4.58
Statistical Analysis 1: Comparison: 15 mg Tirzepatide or MTD vs 4.5 mg Dulaglutide or MTD; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 20.44, 95% CI 2-sided [8.40 to 49.77]

10. Secondary Outcome: Change From Baseline in Fasting Serum Glucose (FSG)
Description: LSMean was calculated using the ANCOVA model for endpoint measures: Variable = Baseline + A1CGR1 + DULDSCRN + OAMGR1 + REGION1 + Treatment (Type I sum of squares).
Time Frame: Baseline, Week 40
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: millimole per liter (mmol/L)
Arm/Group | 15 mg Tirzepatide or MTD | 4.5 mg Dulaglutide or MTD
Number analyzed (Participants) | 123 | 128
millimole per liter (mmol/L) | -2.00 (0.149) | -1.10 (0.150)
Statistical Analysis 1: Comparison: 15 mg Tirzepatide or MTD vs 4.5 mg Dulaglutide or MTD; Test type: Superiority; p < 0.001, ANCOVA; LS Mean difference (Final Values) = -0.90, 95% CI 2-sided [-1.32 to -0.49]

11. Secondary Outcome: Change From Baseline in Waist Circumference
Description: as for outcome 2
Time Frame: Baseline, Week 40
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: centimeter (cm)
Arm/Group | 15 mg Tirzepatide or MTD | 4.5 mg Dulaglutide or MTD
Number analyzed (Participants) | 123 | 111
centimeter (cm) | -8.2 (0.94) | -3.1 (0.97)
Statistical Analysis 1: Comparison: 15 mg Tirzepatide or MTD vs 4.5 mg Dulaglutide or MTD; Test type: Superiority; p = 0.0002, Mixed Models Analysis; LS Mean difference (Final Values) = -5.1, 95% CI 2-sided [-7.8 to -2.5]

12. Secondary Outcome: Change From Baseline in Body Mass Index (BMI)
Description: Change from Baseline in BMI is presented. LSMean was calculated using MMRM for post-baseline measures: Variable = Baseline + Number of Background OAMs Group 1 + Dulaglutide Dose at Screening + Geographic Region 1 + Baseline HbA1c Group + Treatment + Time + Treatment*Time (Type III sum of squares). Variance-Covariance structure (Actual Value) = Unstructured. Variance-Covariance structure (Change from Baseline) = Unstructured.
Time Frame: Baseline, Week 40
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Kilogram per square meter (kg/m^2)
Arm/Group | 15 mg Tirzepatide or MTD | 4.5 mg Dulaglutide or MTD
Number analyzed (Participants) | 123 | 111
Kilogram per square meter (kg/m^2) | -3.9 (0.17) | -1.3 (0.18)
Statistical Analysis 1: Comparison: 15 mg Tirzepatide or MTD vs 4.5 mg Dulaglutide or MTD; Test type: Superiority; p < 0.0001, Mixed Models Analysis; LS Mean difference (Final Values) = -2.6, 95% CI 2-sided [-3.1 to -2.1]

13. Secondary Outcome: Change From Baseline in Impact of Weight on Quality of Life-Lite Clinical Trials Version (IWQOL-Lite CT) - Physical Functioning Score
Description: The IWQOL-Lite-CT is a 20-item, obesity-specific PRO (patient-reported outcome) instrument developed for use in obesity clinical trials. It assesses 2 primary domains of obesity-related health-related quality of life (HRQoL): physical (7 items, where 5 of the items comprise the physical functioning sub-domain) and psychosocial (13 items). The IWQOL-Lite-CT provides composite scores for each domain, as well as a total score, all ranging from 0 to 100. Higher scores reflect better levels of functioning. This endpoint shows results for 'physical function domain.'
Time Frame: Baseline, Week 40
Population: All randomly assigned participants who took at least 1 dose of study drug and had a baseline and at least 1 post-baseline value for this outcome, excluding patients discontinuing study drug due to inadvertent enrollment and data after initiating rescue antihyperglycemic medication or prematurely stopping study drug.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- 4.5 mg Dulaglutide or MTD: Participants received dulaglutide administered as SC injection via a SDP QW for 40 weeks.
  The starting dose of dulaglutide was 0.75 mg QW, which increased by 1.5 mg every 4 weeks (0.75 mg to 1.5 mg to 3 mg to 4.5 mg) until 4.5 mg or MTD was reached.
Arm/Group | 15 mg Tirzepatide or MTD | 4.5 mg Dulaglutide or MTD
Number analyzed (Participants) | 121 | 104
score on a scale | 11.8 (1.77) | 7.8 (1.91)
Statistical Analysis 1: Comparison: 15 mg Tirzepatide or MTD vs 4.5 mg Dulaglutide or MTD; Test type: Superiority; p = 0.1181, ANCOVA; LS Mean difference (Final Values) = 4.1, 95% CI 2-sided [-1.0 to 9.2]

ADVERSE EVENTS:
Time Frame: Baseline up to week 44
Description: All randomized participants who received at least one dose of study drug regardless of adherence to study drug or initiation of rescue medication. Based on the planned safety analysis, adverse events were collected per the treatment regimen, irrespective of each dose level. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Groups:
- 15 mg Tirzepatide or MTD: Participants received 15 mg of tirzepatide administered as SC injection via a SDP QW for 40 weeks.
  The starting dose of tirzepatide was 2.5 mg QW, which increased by 2.5 mg every 4 weeks (2.5 mg to 5 mg to 7.5 mg to 10 mg to 12.5 mg to 15 mg) until 15 mg or MTD was reached.
- 4.5 mg Dulaglutide or MTD: Participants received 4.5 mg of dulaglutide administered as SC injection via a SDP QW for 40 weeks.
  The starting dose of dulaglutide was 0.75 mg QW, which increased by 1.5 mg every 4 weeks (0.75 mg to 1.5 mg to 3 mg to 4.5 mg) until 4.5 mg or MTD was reached.
Arm/Group | 15 mg Tirzepatide or MTD | 4.5 mg Dulaglutide or MTD
All-Cause Mortality (participants affected / at risk) | 1/139 | 1/143
Serious Adverse Events (participants affected / at risk) | 10/139 | 10/143
Other Adverse Events (participants affected / at risk) | 77/139 | 79/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 15 mg Tirzepatide or MTD (N=139) | 4.5 mg Dulaglutide or MTD (N=143)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Dilated cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Microvascular coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Sudden cardiac death (General disorders) | 0 (0) | 1 (1)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/64 (1) | 0/72 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 15 mg Tirzepatide or MTD (N=139) | 4.5 mg Dulaglutide or MTD (N=143)
Abdominal distension (Gastrointestinal disorders) | 7 (8) | 3 (5)
Constipation (Gastrointestinal disorders) | 12 (18) | 11 (17)
Diarrhoea (Gastrointestinal disorders) | 31 (96) | 19 (35)
Dyspepsia (Gastrointestinal disorders) | 11 (26) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 8 (9)
Nausea (Gastrointestinal disorders) | 35 (116) | 27 (62)
Vomiting (Gastrointestinal disorders) | 9 (17) | 14 (34)
Fatigue (General disorders) | 8 (13) | 4 (6)
Covid-19 (Infections and infestations) | 7 (7) | 5 (5)
Influenza (Infections and infestations) | 6 (6) | 14 (15)
Nasopharyngitis (Infections and infestations) | 14 (15) | 12 (17)
Decreased appetite (Metabolism and nutrition disorders) | 12 (14) | 7 (7)
Hyperglycaemia (Metabolism and nutrition disorders) | 5 (5) | 8 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (12) | 4 (4)
Headache (Nervous system disorders) | 8 (12) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-03-09): https://cdn.clinicaltrials.gov/large-docs/39/NCT05564039/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-01): https://cdn.clinicaltrials.gov/large-docs/39/NCT05564039/SAP_001.pdf